CLINICAL TRIAL: NCT06848387
Title: Concentration of Unbound Cloxacillin in Adults Treated With Continuous Infusion Via Elastomeric Pump
Brief Title: Unbound Cloxacillin Concentrations During Continuous Infusion
Acronym: KLONC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emeli Månsson (Other)
Collaborators: Region Västmanland (Other)
Responsible Party: Sponsor-Investigator, Emeli Månsson, Principal Investigator, Region Västmanland
Organization: Region Västmanland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 992496/KLONC
Record Dates: First submitted 2025-01-15; First posted 2025-02-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Staphylococcal Infections
Keywords: cloxacillin
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Low intervention trial according to Regulation (EU) No 536/2014. The investigational medical product - cloxacillin - is authorized and according to the protocol of the clinical trial
  1. Cloxacillin is used in accordance with the terms of the marketing authorization
  2. The use of cloxacillin is evidence-based
  3. The additional monitoring procedures - four blood samples drawn before, after 4h, after 24h, and after 48h of continuous infusion of cloxacillin - do not pose more than minimal additional risk or burden to the safety of the subjects compared to normal clinical practice.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with cloxacillin as continuous infusion via elastomeric pump (Experimental): Additional monitoring procedures performed: blood samples drawn before, after 4h, after 24h, and after 48h of continuous infusion of cloxacillin.
  Interventions: Diagnostic Test: Unbound cloxacillin concentration

INTERVENTIONS:
Diagnostic Test: Unbound cloxacillin concentration — Unbound cloxacillin concentration measured at baseline, after 4h, after 24h and after 48h of continuous infusion.

SUMMARY:
Cloxacillin is the first-line choice for the treatment of severe infections caused by the bacterium Staphylococcus aureus in Sweden. Over the past year, cloxacillin is increasingly administred through continuous infusion. In this study, the free (unbound) concentration of cloxacillin when administered as a continuous infusion will be measured to ensure that the free concentration is neither too high nor too low. A PK/PD model will be developed to predict which dosage of cloxacillin is appropriate for an individual based on age, gender, kidney function, and serum-protein level.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Treating physician has decided to start continuous infusion of cloxacillin

Exclusion Criteria:

* Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Free (unbound) cloxacillin concentration | From enrollment to end of follow up at 48 hours

IPD SHARING:
Plan to Share IPD: No